CLINICAL TRIAL: NCT01607203
Title: Randomised Controlled Trial Comparing hCG Triggering Versus hCG Associated With GnRH Agonist
Brief Title: Trial Comparing hCG Triggering Versus hCG Associated With GnRH Agonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Jan Palfijn Gent (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Dr. Decleer Wim, gynaecologist, AZ Jan Palfijn Gent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr. Decleer Wim
Record Dates: First submitted 2012-05-04; First posted 2012-05-30 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Infertility
Keywords: ovarian hyper stimulation syndrome (OHSS); metaphase II oocytes (MII); good quality embryo's; implantation; pregnancy
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hCG (Active Comparator): 5000 IU Pregnyl SC
  Interventions: Drug: pregnyl
- hCG and GnRH agonist (Active Comparator): 5000 IU Pregnyl SC + 0.2 mg Decapeptyl daily SC
  Interventions: Drug: Decapeptyl Daily; Drug: pregnyl

INTERVENTIONS:
Drug: Decapeptyl Daily — Decapeptyl 0.2 mg SC once 1day
  Other Names: Gonapeptyl
  Arms: hCG and GnRH agonist
Drug: pregnyl — 5000 IU SC

SUMMARY:
The purpose of this study is to see whether patients triggered with only human Chorion Gonadotropin (hCG) have higher number of Metaphase II oocytes (MII) and implantation rate than patients triggered with hCG combined with Gonadotropin Releasing Hormone (GnRH) agonist.

ELIGIBILITY:
Inclusion Criteria:

* Intra-cytoplasmic sperm injection (ICSI) patients below 38 years
* 1,2 or 3 rd IVF-cycle

Exclusion Criteria:

* polycystic ovary syndrome (PCOS) patients
* patients with endocrinological diseases or problems

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Decleer, gynacologist, Principal Investigator — IVF Centrum Jan Palfijn Gent
Locations (1):
- A Z Jan Palfijn, Ghent, Oost-vlaanderen, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: the Principal Investigator (PI) prescreened the patients and only the eligible patients were assigned to a group by the study coordinator
Groups:
- hCG Triggering: TRIGGERING FOR FINAL MATURATION BY 5000 IU PREGNYL SC ONLY 36 HOURS BEFORE OOCYTE RETRIEVAL
- hCG and GnRH Agonist Triggering: DUAL TRIGGERING FOR FINAL MATURATION BY 5000IU PREGNYL SC AND DECAPEPTYL(GONAPEPTYL) 0.2 MG SC 36 HOURS BEFORE OOCYTE RETRIEVAL
Period: Overall Study
Arm/Group | hCG Triggering | hCG and GnRH Agonist Triggering
Started | 59 | 61
Completed | 59 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCG TRIGGERING | hCG and GnRH Agonist Triggering | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 30.5 (4.1) | 30.0 (3.6) | 30.2 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants] — FEMALE
  Participants
    Female | 59 | 61 | 120
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 59 | 61 | 120
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (5.1) | 23.8 (4.6) | 23.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: MII Oocytes
Description: the number of mature oocytes retrieved
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: cumulus oocyte complex
Arm/Group | hCG TRIGGERING | hCG and GnRH Agonist Triggering
Number analyzed (Participants) | 59 | 61
cumulus oocyte complex | 9.2 (6.7) | 10.3 (6.8)

2. Secondary Outcome: Pregnancy Rate
Description: the number of pregnancies obtained, wich still is the most important issue for the patients
Time Frame: 12 weeks
Measure: Number; unit: pregnancies
Arm/Group | hCG Triggering | hCG and GnRH Agonist Triggering
Number analyzed (Participants) | 59 | 61
pregnancies | 28 | 45

3. Secondary Outcome: Patients With Cryopreserved Embryos
Time Frame: 4 weeks
Measure: Number; unit: patients with cryopreserved embryos
Arm/Group | hCG Triggering | hCG and GnRH Agonist Triggering
Number analyzed (Participants) | 59 | 61
patients with cryopreserved embryos | 21 | 33
Statistical Analysis 1: Comparison: hCG Triggering vs hCG and GnRH Agonist Triggering; Test type: Non-Inferiority or Equivalence — t -test; p = 0.04, Fisher Exact

ADVERSE EVENTS:
Arm/Group | hCG TRIGGERING | hCG and GnRH Agonist Triggering
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCG TRIGGERING (N=59) | hCG and GnRH Agonist Triggering (N=61)
OHSS (Metabolism and nutrition disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No